CLINICAL TRIAL: NCT02434172
Title: The CryptoART Study: Decreasing Mortality Associated With Initiation of Antiretroviral Therapy in Sub-Saharan Africa Through Early Detection and Prevention of Cryptococcal Disease
Brief Title: CryptoART Study: Decreasing Mortality Associated With Initiation of Antiretroviral Therapy in Sub-Saharan Africa
Acronym: CryptoART
Status: Completed | Type: Observational
Sponsor: University of Zimbabwe (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chiratidzo Ndhlovu, Associate Professor of Medicine, University of Zimbabwe
Other Study IDs: 1U01GH000737-01 (NIH)
Record Dates: First submitted 2015-04-24; First posted 2015-05-05 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Cryptococcal Meningitis
Keywords: HIV; Cryptococcus; Lateral Flow Assay; sub-Saharan Africa; Screening; treatment; cryptococcal meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, and peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Screening: There are no arms to the study. All participants will undergo screening. Preemptive treatment will only be provided to those who are CrAg positive.
  Interventions: Other: Pre-emptive screening and treatment for cryptococcal disease

INTERVENTIONS:
Other: Pre-emptive screening and treatment for cryptococcal disease — Preemptive screening for cryptococcal disease among individuals with CD4 counts below 100 cells/mm3 with anti fungal therapy for those what are Cryptococcus antigen positive. These participants will be followed longitudinally for 12 months to determine clinical outcome, with their outcome compared with similar patients who are cryptococcal antigen negative, who will also be followed longitudinally for 12 months.

SUMMARY:
The study will determine if the initiation of a 'screen and treat' program for cryptococcal disease among HIV positive individuals decreases morbidity and mortality among individuals with CD4 count < 100 cells/mm3. The study will screen individuals who are asymptomatic for CM and are either ART naïve or ART experienced with CD4 count < 100 cells/mm3.

The introduction of an cheap, easy to use point of care diagnostic test the lateral flow assay will facilitate rapid diagnosis of cryptococcal disease in resource limited settings. The investigators will determine the efficacy of the lateral flow assay in identifying latent and asymptomatic cryptococcal disease. The investigators will determine the efficacy of the test in detecting disease in readily available body fluids such as urine and whole blood obtained via finger-stick method. The investigators will also determine the cost effectiveness of a screen and treat approach for cryptococcal disease in Zimbabwe.

The investigators also wish to understand why some individuals with low CD4 counts reactivate cryptococcal disease and screen positive for cryptococcal antigen (CrAg) while others with similar levels of immunocompromised do not.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV positive test by standard national algorithm
* CD4 count ≤100 cells/mm3
* Age > 18 years
* Residence within 50 km of Harare
* Able to provide written informed consent

Exclusion Criteria:

* Presence of clinical symptoms suggestive of meningitis.
* Recent history of CM within 2 weeks of enrollment, i.e., participants within the induction phase of therapy.
* Individuals with severe hepatic injury, jaundice, alanine transferase (ALT) >5x upper limit of normal
* Individuals with renal failure, defined by an estimated Glomerular filtration rate (eGFR) ≤30 mL/min (using MDRD (Modification of Diet in Renal Disease) equation)
* Currently known to be pregnant
* A negative urine pregnancy test is required for study entry for women with childbearing potential.
* The use of contraception will be recommended to women with childbearing potential while on high dose fluconazole therapy. Referral to family planning services will be given as necessary.
* Previous allergy or other reaction to amphotericin B and/or fluconazole
* Currently enrolled in another clinical trial/study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit Asymptomatic participants with severe immunosuppression at risk of cryptococcal disease. The individuals will have a CD4 count <100cells/mm3 and can be ART naive or ART experienced with no symptoms of active Cryptococcal disease.
  They will be recruited from outpatient HIV/ART clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1333 (Actual)
Dates: Start 2015-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
12- month survival in CrAg-positive persons vs. CrAg-negative persons screened | 12 months

SECONDARY OUTCOMES:
Seroprevalence of asymptomatic cryptococcal antigenemia among individuals with CD4≤100 cells/mm3 in an urban population in Zimbabwe | 24 months
Sensitivity, specificity, positive and negative predictive values of point-of-care urine CrAg LFAs | 24 months
Sensitivity, specificity, positive and negative predictive values of point-of-care whole blood CrAg LFAs | 24 months
Proportion of individuals with CD4≤100 cells/mm3 and a positive CrAg assay who have disseminated cryptococcal infection with either blood infection or CSF involvement | 24 months
12-month survival among individuals with CD4≤100 cells/mm3 prior to implementation of CrAg screening program using historical controls | 24 months
  Retrospective analysis
Cost of implementation of CrAg screening among individuals with CD4≤100 cells/mm3 | 24 months
Cryptococcus-associated mortality among individuals with CD4≤100 cells/mm3, | 24 months
Incidence of cryptococcal and non-cryptococcal IRIS | 24 months
Barriers to uptake of diagnostic LP by individuals with asymptomatic cryptococcal antigenemia. | 24 months
  Questionnaire will be administered to participants who are serum cryptococcal antigen positive who decline to undergo LP.
Inflammatory cytokines and functional impairments in antigen specific T cells that are associated with the development of cryptococcal antigenemia and meningitis. | 24 months
  Analysis will be done by ELISA and Luminex assays, cell culture and flow cytometry techniques, data collected will be entered into a database and analyzed by patient characteristics.
Impact of ART mediated immune reconstitution on the inflammatory cytokine profile and the cryptococcal antigen specific CD4+ T cell response in those with serum and CSF cryptococcal antigenemia compared with those without. | 24 months
  Analysis will be done by ELISA and Luminex assays, cell culture and flow cytometry techniques, data collected will be entered into a database and analyzed by patient characteristics. Data will be longitudinal including baseline characteristics and subsequent follow-up data at 6 months and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Chiratidzo E Ndhlovu, MBBS, MSc, Principal Investigator — University of Zimbabwe College of Health Sciences; Azure T Makadzange, MD DPhil, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Parirenyatwa Hospital, Harare, Zimbabwe

REFERENCES:
- [Derived] Kouamou V, Gundidza P, Ndhlovu CE, Makadzange AT; CryptoART Study Team. Effects of Gender and Baseline CD4 Count on Post-Treatment CD4 Count Recovery and Outcomes in Patients with Advanced HIV Disease: A Retrospective Cohort Study. AIDS Res Hum Retroviruses. 2023 Jul;39(7):340-349. doi: 10.1089/AID.2022.0117. Epub 2023 Apr 26. PMID 36924288
- [Derived] Boyd K, Kouamou V, Hlupeni A, Tangwena Z, Ndhlovu CE, Makadzange AT; CryptoART Study Team. Diagnostic Accuracy of Point of Care Cryptococcal Antigen Lateral Flow Assay in Fingerprick Whole Blood and Urine Samples for the Detection of Asymptomatic Cryptococcal Disease in Patients with Advanced HIV Disease. Microbiol Spectr. 2022 Aug 31;10(4):e0107522. doi: 10.1128/spectrum.01075-22. Epub 2022 Aug 4. PMID 35924841